CLINICAL TRIAL: NCT01263912
Title: Essential Fatty Acid Nutrition in Infants 1 to 2 Years-of-Age
Brief Title: Essential Fatty Acid Nutrition For 1-2 Yr-Olds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry); DSM Food Specialties (Industry)
Responsible Party: Principal Investigator, Angela Devlin, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: H09-02028
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Infant Nutrition
Keywords: Polyunsaturated fatty acids; Cognitive development; Growth; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCPUFA Supplement (Active Comparator): DHA/ARA supplement providing 200 mg/day docosahexaenoic acid (DHA) from DHASCO®-S oil and 200 mg/day arachidonic acid (ARA) from ARASCO® oil (DSM Nutritional Products).
  Interventions: Dietary Supplement: LCPUFA Supplement
- A Placebo (Placebo Comparator): 400 mg/day corn oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: LCPUFA Supplement — Children 12-13 months old will be assigned at random to receive either a nutrition supplement containing LCPUFA or a placebo until 24 months-of-age
  Arms: LCPUFA Supplement
Dietary Supplement: Placebo — Children 12-13 months old will be assigned at random to receive either a nutrition supplement containing LCPUFA or a placebo until 24 months-of-age
  Arms: A Placebo

SUMMARY:
This is a prospective longitudinal study that will involve 200 infants enrolled at 12-13 months of age. The study will use a classic nutrition design to assess if infants' feeding practices in Canada place infants 1-2 years of age at risk for low long chain polyunsaturated fatty acid (LCPUFA), nutrients known to influence growth, and brain and immune system development. On enrollment, infants will be assigned at random to a nutrition supplement providing omega 6 and omega 3 LCPUFA or a PUFA placebo.

DETAILED DESCRIPTION:
The objectives are to1. determine the change in dietary fat and PUFA intakes, change in biochemical measures of fatty acid status prospectively from enrollment to 24 months-of-age and 2. to use a nutritional intervention with LCPUFA to address if limiting status of these nutrients impacts growth and development to 24 months-of-age. Primary Endpoints are distributions of developmental tests scores, growth quality and parental reports of child illness. The Bayley Mental and Motor Scales (BSID-III), Peabody Picture Test, Beery Buktenica Developmental Test, Auditory Continuous Performance Test and Test of Attention and Distractibility are used. Growth is assessed as height, weight, and adipose tissue mass and distribution. Child illness is reported by the parent. Secondary endpoints are physiologic measures of blood pressure, heart rate and heart rate variability, and the genetic variables in fatty acid metabolism on fatty acid status and outcome. Blood is collected at enrolment and at 24 months-of-age. Lipids and fatty acids are assessed on plasma and blood cells. Routine, potentially confounding nutrients including iron, vitamin D, choline, folate and B12 are assessed. DNA is extracted from blood cells for genotyping. Dietary intake is assessed using a food frequency questionnaire (FFQ), 3 day food diaries and 24 hour recalls. A parent report illness dairy and questionnaire modified from the International Study of Asthma and Allergies in Childhood is used to assess illness incidence and duration. Descriptive statistics will be used to present subject characteristics, dietary intakes, growth and physiological measures and test results of total fat. Logistic regression, with multivariable-adjusted odds ratios (ORs) of a negative outcome and corresponding 95% CI will be sued to assess the effect of LCPUFA status on development, growth and health outcomes. For all multivariate models, potential confounders will be screened in stepwise fashion, and any covariate with a regression coefficient P-value < 0.05 (two-sided) will be retained. Performance on tests will be compared as LCPUFA status in the lowest quintile compared to highest quintile of outcome (i.e. the two ends of the distribution differ in LCPUFA status).

ELIGIBILITY:
Inclusion criteria:

* term gestation (37-41 weeks gestation and 2500g or more at birth)
* single birth
* English as the primary language in the home
* non-smoking home environment
* a healthy infant not yet 13 months-of-age, who is not currently breast-fed or fed infant formula with ARA and DHA.
* primary milk source is cows' milk, cows' milk substitutes, or other milk substitutes containing no supplemental fatty acids from enrollment to 24 months-of age.
* the infant has no known food allergies, metabolic, neurological, genetic, or immune disorders that are likely, in the opinion of the investigator to impact the outcome measures in this study.
* the infant has not been fatty acid or oil, including fish oil supplements and there is no intent to provide these supplements during the study.
* the infant has no history of hospitalization, growth failure or any other event which in the opinion of the investigator is likely to impact the outcome measures in this study.

Exclusion Criteria:

* any infant that does not meet the inclusion criteria will not be included in this study.

Ages: 12 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2010-12; Primary Completion 2015-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Developmental test scores | 12 months (at 24 months of age)
  Bayley Scales of Infant and Toddler Development 3rd Edition and Beery-Buktenica Developmental Test of Visual -Motor Integration (5th Ed) composite scores at 24 months in relation to LCPUFA supplement group.

SECONDARY OUTCOMES:
Plasma and Red Blood Cell fatty acids (% total fatty acids) | 12 months (at 24 months of age)
  Plasma and red blood cell fatty acids levels in relation to dietary LCPUFA intake
Systolic and diastolic blood pressure (mmHg) | 12 months (at baseline and 24 months of age)
  In clinic systolic and diastolic blood pressure in relation to LCPUFA status
Heart rate and heart rate variability | 12 months (at baseline and 24 months of age)
  Heart rate and heart rate variability in relation to LCPUFA status
Genetic variation in fatty acid desaturases | 12 months (at 24 months of age)
  Genetic variation in fatty acid desaturases in relation to LCPUFA status
Hemoglobin (g/dL) | 12 months (at baseline and 24 months of age)
  Hemoglobin concentration in relation to diet
Ferritin (ng/ml) | 12 months (at baseline and 24 months of age)
  Serum ferritin in relation to child diet
Choline metabolites (umol/L) | 12 months (at baseline and 24 months of age)
  Plasma free choline, betaine, and dimethylglycine in relation to child diet
Folate (nmol/L) | 12 months (at baseline and 24 months of age)
  Serum folate in relation to child diet
Vitamin B12 (pmol/L) | 12 months (at baseline and 24 months of age)
  Serum vitamin B12 in relation to child diet
Vitamin D (nmol/L) | 12 months (at baseline and 24 months of age)
  Serum vitamin D in relation to child diet
Supplements and supplemented foods | 12 months (at baseline and age 18 and 24 months)
  Use of nutrient supplements and supplemented foods and child nutrient status.
Growth (weight, kg) | 12 months (at baseline and age 18 and 24 months)
  Weight of at baseline, 18 and 24 months in relation to LCPUFA
Growth (height) | 12 months (at baseline and age 18 and 24 months)
  Height at baseline, 18 and 24 months in relation to LCPUFA
Growth (BMI, kg/m2) | 12 months (at baseline and age 18 and 24 months)
  BMI at baseline, 18 and 24 months in relation to LCPUFA
Growth (waist circumference, cm) | 12 months (at baseline and age 18 and 24 months)
  Waist circumference at baseline, 18 and 24 months in relation to LCPUFA
Incidence and duration of illness | 12 months (at baseline and age 18 and 24 months)
  Parental reports of illness and duration

CONTACTS AND LOCATIONS:
Overall Officials: Angela Devlin, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Devlin AM, Chau CMY, Dyer R, Matheson J, McCarthy D, Yurko-Mauro K, Innis SM, Grunau RE. Developmental Outcomes at 24 Months of Age in Toddlers Supplemented with Arachidonic Acid and Docosahexaenoic Acid: Results of a Double Blind Randomized, Controlled Trial. Nutrients. 2017 Sep 6;9(9):975. doi: 10.3390/nu9090975. PMID 28878181
- [Derived] Wiedeman AM, Dyer RA, McCarthy D, Yurko-Mauro K, Innis SM, Devlin AM. Biomarkers of Docosahexaenoic Acid but Not Arachidonic Acid Reflect Dietary Intakes in Toddlers at Ages 1 and 2 Years Who Are Not Meeting Dietary Recommendations. J Nutr. 2020 Mar 1;150(3):518-525. doi: 10.1093/jn/nxz280. PMID 31754697
- [Derived] Wiedeman AM, Chau CMY, Grunau RE, McCarthy D, Yurko-Mauro K, Dyer RA, Innis SM, Devlin AM. Plasma Betaine Is Positively Associated with Developmental Outcomes in Healthy Toddlers at Age 2 Years Who Are Not Meeting the Recommended Adequate Intake for Dietary Choline. J Nutr. 2018 Aug 1;148(8):1309-1314. doi: 10.1093/jn/nxy108. PMID 29986040